CLINICAL TRIAL: NCT01509495
Title: Impedance Measurements in Heart Failure Patients
Acronym: SIM-HF
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Enrollment rate too low; rate much under estimation of sponsor and investigators
Sponsor: Medtronic BRC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RAE00564
Record Dates: First submitted 2011-12-07; First posted 2012-01-13 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-05

CONDITIONS: Heart Failure
Keywords: Heart Failure; HF
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Akern BIA101 and Custom Device — Impedance Measurement every 4 hours

SUMMARY:
The purpose of this study is to measure impedance during inpatient treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to hospital for symptoms of congestive heart failure
* patients older than 18 years
* patients willing and able to give informed consent

Exclusion Criteria:

* patients who will require adrenergic or positive inotropic medications
* patients enrolled in a concurrent study that may confound the results of this study
* patients unable or unwilling to participate in study procedures
* patients who are pregnant
* patients who are mentally handicapped or legal incompetent
* patients who are dependent on investigator or sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Impedance Measurement of Patients in Heart Failure, impedance change first to last measurement | every 4 hours up to 48 hours

SECONDARY OUTCOMES:
Accuracy of Respiratory rate determined by impedance measurements | every 4 hours up to 48 hours
Correlation between hemodynamic (central venous or arterial pressure) and impedance measurements (optional) | every 4 hours up to 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian KG Maier, Prof., Principal Investigator — Klinikum St. Elisabeth Straubing, Med. Klinik II, St.-Elisabeth-Str. 23, 94315 Straubing, Germany; Eva Goncalvesova, Prof., Principal Investigator — NUSCH, Cardiac Surgery, Pod Krasnou horkou 1, 83348 Bratislava, Slovakia; Petr Neuzil, Prof., Principal Investigator — Nemocnice Na Homolce, Cardiology, Roentgenova 2/37, 150 30 Praha 5, Czechia
Locations (3):
- Nemocnice Na Homolce, Prague, Czechia
- Universitätsklinik Würzburg, Medizinische Klinik und Poliklinik I, Würzburg, Franken, Germany
- NUSCH, Bratislava, Slovakia